CLINICAL TRIAL: NCT00580645
Title: Do Treatments for Smoking Cessation Affect Alcohol Drinking?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sherry McKee, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIC0702002391; R01AA015596-01 (NIH)
Record Dates: First submitted 2007-12-25; First posted 2007-12-27 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Alcohol Drinking
Keywords: alcohol; smoking cessation; varenicline; bupropion; smoking cessation medications
MeSH Terms: conditions — Alcohol Drinking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Experimental): varenicline 1mg/day or 2mg/day
  Interventions: Drug: varenicline
- Placebo (Placebo Comparator): Placebo Controlled
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — 2mg/day or 1mg/day with 1-week medication lead-in period.
  Other Names: Chantix
  Arms: varenicline
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of smoking cessation medications on alcohol drinking. Effect of 2mg/day, 1mg/day, placebo varenicline was evaluated.

Following 7 days of medication pre-treatment to achieve steady state levels, participants complete a laboratory session assessing alcohol self-administration behavior.

Study enrolls heavy drinking smokers (not tested under nicotine deprivation), non-daily smokers, and nonsmokers. Volunteers are administered either varenicline (Chantix) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or older
* Able to read and write in English
* Smokers, non-daily smokers, and non-smokers
* Heavy Drinkers and/or meet criteria for alcohol use disorders

Exclusion Criteria:

* Any significant current medical or psychiatric conditions that would contraindicate the consumption of alcohol
* Significant hepatocellular injury
* Positive test result at intake appointments on urine drug screens conducted for opiates, cocaine, or benzodiazepines
* Women who are pregnant or nursing
* Suicidal, homicidal, or evidence of severe mental illness
* Prescription of any psychotropic drug in the 30 days prior to study enrollment
* Blood donation within the past 8 weeks
* Individuals who are seeking treatment for drinking or smoking or who have attempted to quit drinking or smoking within the past 3 months
* Specific exclusions for administration of bupropion not specified above including: having taken monoamine inhibitors in the past six weeks; history of anorexia or bulimia; previous hypersensitivity to bupropion; history of alcohol or drug dependence in the past year; history of seizure disorder of any etiology
* Known allergy to varenicline or taking H2blockers
* Participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current study
* Subjects likely to exhibit clinically significant alcohol withdrawal during the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation and Yale Behavioral Pharmacology Laboratory, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Roberts W, McKee SA. Effects of varenicline on cognitive performance in heavy drinkers: Dose-response effects and associations with drinking outcomes. Exp Clin Psychopharmacol. 2018 Feb;26(1):49-57. doi: 10.1037/pha0000161. PMID 29389170

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 mg/Day Varenicline: 1mg/day with 1-week medication lead-in period. The starting dose is 0.5 mg/day for days 1-5, followed by 0.5mg twice daily for days 6-7. 0.5mg twice daily administered during laboratory session (day 8) and for 4 weeks after laboratory session.
- 2 mg/Day Varenicline: 2mg/day with 1-week medication lead-in period. The starting dose is 0.5 mg/day for Day 1 and 2, 0.5 mg twice daily for Days 3-5, and 1.0mg twice daily on Days 6-7. 1.0mg twice daily administered during laboratory session (day 8) and for 4 weeks after laboratory session.
Period: Overall Study
Arm/Group | Placebo | 1 mg/Day Varenicline | 2 mg/Day Varenicline
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 1 mg/Day Varenicline | 2 mg/Day Varenicline | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (9.52) | 33.35 (8.51) | 34.15 (11.6) | 33.90 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 5 | 19
  Male | 14 | 12 | 15 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 1 | 1 | 2
  African American | 8 | 7 | 2 | 17
  White | 11 | 10 | 15 | 36
  Other | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Consumed
Description: number of drinks consumed during hour 1 and hour 2 of the 120 minute alcohol self-administration session
Time Frame: 2 hour ad-lib drinking period, during the laboratory session (Day 8)
Population: number of drinks consumed during hour 1 and hour 2 of the 120 minute alcohol self-administration session
Measure: Mean (Standard Error); unit: number of drinks
Arm/Group | Placebo | 1 mg/Day Varenicline | 2 mg/Day Varenicline
Number analyzed (Participants) | 20 | 20 | 20
number of drinks
  hour 1 | 2.1 (0.37) | 2.05 (0.32) | 1.5 (0.33)
  hour 2 | 1.7 (0.37) | 2.05 (0.37) | 1.5 (0.37)

2. Secondary Outcome: Alcohol Craving
Description: alcohol craving during the alcohol priming dose period using a visual analog scale of alcohol craving (1-100; higher scores = higher craving)
Time Frame: during laboratory session (Day 8) at baseline
Population: n=19 in the 2mg/day varenicline group because 1 subject failed to respond on measure.
Measure: Mean (Standard Error); unit: units on a visual analog scale
Arm/Group | Placebo | 1 mg/Day Varenicline | 2 mg/Day Varenicline
Number analyzed (Participants) | 20 | 20 | 19
units on a visual analog scale | 37.24 (5.32) | 34.11 (5.32) | 24.04 (5.33)

ADVERSE EVENTS:
Time Frame: Titration period (8 days).
Description: All adverse events reported during 1 week medication period. Baseline reporting not controlled. Subjects were queried about the presence/absence of severity of common symptoms (>5% from placebo according to manufacturer) associated with varenicline. Adverse events assessed on Day 1, 2, 5, and Day 8.
Arm/Group | Placebo | 1 mg/Day Varenicline | 2 mg/Day Varenicline
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 4/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | 1 mg/Day Varenicline (N=20) | 2 mg/Day Varenicline (N=20)
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 6 | 4 | 5
Dry Mouth (General disorders) | 7 | 2 | 2
Insomnia (General disorders) | 2 | 0 | 5
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Difficulty Breathing (General disorders) | 0 | 1 | 1
Shortness of Breath (General disorders) | 1 | 0 | 1
Tightness in Chest (Cardiac disorders) | 0 | 1 | 0
Abnormal Dreams (General disorders) | 2 | 1 | 3
Fast Heartbeat (Cardiac disorders) | 1 | 1 | 3
Suicidal Thoughts (General disorders) | 0 | 0 | 0
Erratic Behavior (General disorders) | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No